CLINICAL TRIAL: NCT04361552
Title: Tociluzumab for Cytokine Release Syndrome With SARS-CoV-2: An Open-Labeled, Randomized Phase 3 Trial
Brief Title: Tocilizumab for the Treatment of Cytokine Release Syndrome in Patients With COVID-19 (SARS-CoV-2 Infection)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study abandoned due to drug billing issues
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000419; NCI-2020-02314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP4998-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-24 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Cerebrovascular Accident; Chronic Obstructive Pulmonary Disease; Chronic Renal Failure; Coronary Artery Disease; Diabetes Mellitus; Malignant Neoplasm; SARS Coronavirus 2 Infection
MeSH Terms: conditions — Stroke; Pulmonary Disease, Chronic Obstructive; Kidney Failure, Chronic; Coronary Artery Disease; Diabetes Mellitus; Neoplasms; COVID-19 | interventions — Practice Guidelines as Topic; Standard of Care; tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (tocilizumab, standard of care) (Experimental): Patients receive tocilizumab IV every 12 hours for up to 3 doses in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care.
  Interventions: Other: Best Practice; Biological: Tocilizumab
- Arm II (standard of care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Biological: Tocilizumab — Given IV
  Other Names: Actemra; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA; R-1569; RoActemra
  Arms: Arm I (tocilizumab, standard of care)

SUMMARY:
This phase III trial compares the effect of adding tocilizumab to standard of care versus standard of care alone in treating cytokine release syndrome (CRS) in patients with SARS-CoV-2 infection. CRS is a potentially serious disorder caused by the release of an excessive amount of substance that is made by cells of the immune system (cytokines) as a response to viral infection. Tocilizumab is used to decrease the body's immune response. Adding tocilizumab to standard of care may work better in treating CRS in patients with SARS-CoV-2 infection compared to standard of care alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To decrease the length of invasive mechanical ventilation (MV) and rate of 30-day mortality from CRS due to SARS-CoV-2.

SECONDARY OBJECTIVES:

I. To decrease the rates of intensive care unit (ICU) transfer. II. To decrease the rate of invasive mechanical ventilation (MV). III. To decrease the length of ICU stay. IV. To decrease the rate of tracheostomy. V. Safety and efficacy of tociluzumab. VI. Biomarker assessment for response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive tocilizumab intravenously (IV) every 12 hours for up to 3 doses in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care.

ARM II: Patients receive standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with SARS-CoV-2 by the currently available assays (Food and Drug Administration [FDA] approved)
* Should be hospitalized and exhibit at least one of the following predictors of mortality

  * Age >= 65 years
  * Current smoker (smoked >= 100 cigarettes in life and actively smoking)
  * Chronic obstructive pulmonary disease (COPD)
  * Diabetes
  * Hypertension
  * Coronary artery disease
  * Cerebrovascular accident (CVA)
  * Chronic renal disease (creatinine of >= 2 mg/dl)
  * Cancer
  * Patients that have C-reactive protein (CRP) >= 10 mg/L
  * D-dimer >= 0.5 mg/L
  * Procalcitonin >= 0.5 mg/L
  * Lactate dehydrogenase (LDH) >= upper limit of normal (ULN)
* Patients or authorized family member willing to sign informed consent to participate in this study

Exclusion Criteria:

* Pregnant or lactating women
* Hypersensitivity to tocilizumab
* Patients or authorized family member unwilling to sign informed consent to participate in this study
* Uncontrolled tuberculosis, or any uncontrolled fungal infection (eg: candidemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
7-day length of invasive mechanical ventilation (MV) | Up to 7 days
  The 7-day length of invasive MV for each arm will be estimated with 95% confidence intervals (CIs) using the exact binomial distribution. Their difference by the arms will be tested by Cochran-Mantel-Haenszel (CMH) test stratified by the age group and Sequential Organ Failure Assessment (SOFA) score at significance level of 0.05.
30-day mortality rate | Up to 30-day after randomization
  Defined as death within 30-day after randomization. The 30-day mortality rate for each arm will be estimated with 95% CIs using the exact binomial distribution. Their difference by the arms will be tested CMH test stratified by the age group and SOFA score at significance level of 0.05.

SECONDARY OUTCOMES:
Rate of intensive care (ICU) transfer | Up to 2 years
  The rate of ICU transfer for each arm will be estimated with 95% CIs using the exact binomial distribution. Their difference by the arms will be tested CMH test stratified by the age group and SOFA score at significance level of 0.05.
Rate of invasive mechanical ventilation | Up to 2 years
  The rate of invasive mechanical ventilation for each arm will be estimated with 95% CIs using the exact binomial distribution. Their difference by the arms will be tested CMH test stratified by the age group and SOFA score at significance level of 0.05.
Rate of tracheostomy | Up to 2 years
  The rate of tracheostomy for each arm will be estimated with 95% CIs using the exact binomial distribution. Their difference by the arms will be tested CMH test stratified by the age group and SOFA score at significance level of 0.05.
Length of ICU stay | Up to 2 years
  Will first be described by median and inter-quartile, and then compared between two arms by Wilcoxon Sum-Rank test
Length of hospital stay | Up 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Nooka, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.